CLINICAL TRIAL: NCT00577395
Title: A 12-month, Multicenter, Double-blind, Randomized, Parallel Group Study Comparing 150 mg Once-a-month Risedronate and Placebo Using 3-dimensional Micro MRI (Magnetic Resonance Imaging).
Brief Title: Bone Microarchitecture in Osteopenic Postmenopausal Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007075
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): one 150 mg risedronate once a month, orally
  Interventions: Drug: risedronate
- 1 (Placebo Comparator): Placebo tablet once a month, orally
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — oral tablet once a month for 12 months
  Arms: 1
Drug: risedronate — tablet, 150 mg once a month for 12 months
  Arms: 2

SUMMARY:
The purpose of this trial is to compare the difference in bone microarchitecture of the distal radius at month 12 in postmenopausal osteopenic women treated with risedronate 150mg taken once a month compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female: 40 and 57 years of age inclusive
* cessation of menstruation (surgical or natural) between 12 and 36 months prior to study enrollment
* have osteopenia defines as having the following: have osteopenia defined as having the following:
* Lumbar spine (L1-L4) Bone Mineral Density (BMD) T score -1 and less than -2.5 AND a total hip T score of greater than -2.5 OR
* Lumbar spine (L1-L4) BMD T score greater than -2.5 AND a total hip T score -1 and less than -2.5;
* have a body mass index (BMI) between 18 and 30 kg/m2.

Exclusion Criteria:

* history of uncontrolled hyperparathyroidism, hyperthyroidism, osteomalacia
* use of medications within 3 months of starting study drug that impact bone metabolism such as glucocorticoids, estrogens, calcitonin, calcitriol, other bisphosphonates and parathyroid hormone
* hypocalcemia or hypercalcemia of any cause

Ages: 40 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Balske, MD, PhD, Study Director — Procter and Gamble
Locations (4):
- United States (3):
  - Research Facility, Tuscon, Arizona
  - Research Facility, Omaha, Nebraska
  - Research Site, Cincinnati, Ohio
- Research Facility, Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning with the first patient screened on June 18th, 2008, a total of 51 patients were screened for inclusion into the study, of which 38 were excluded from further participation.
Pre-assignment Details: The Screening visit was conducted within 45 days of randomization. After obtaining written informed consent, patients underwent a preliminary screening, including Dual Energy X-ray Absorptiometry (DXA) of the lumbar spine and proximal femur. The most frequent reason for screening failure was DXA results.
Groups:
- One 150 mg Risedronate Once a Month: one 150 mg risedronate once a month, orally
- Placebo Tablet Once a Month: Placebo tablet once a month, orally
Period: Overall Study
Arm/Group | One 150 mg Risedronate Once a Month | Placebo Tablet Once a Month
Started | 7 (67 planned for Treatment 2, but due to enrollment difficulties this was not met.) | 6 (67 were planned for Treatment 1, but due to enrollment difficulties this was not met.)
Completed | 0 (The study was terminated early by the Sponsor for lack of enrollment) | 0 (The study was terminated early by the Sponsor for lack of enrollment)
Not Completed | 7 | 6
Not completed — Study was terminated early by Sponsor | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One 150 mg Risedronate Once a Month | Placebo Tablet Once a Month | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 51.42 (2.50) | 53.83 (2.63) | 52.53 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
  Argentina | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Erosion Index (A Ratio of Curve-like Structures to Plate-like Structures and is a Measure of the Degree of Structural Degradation) of the Distal Radius
Description: The percent was change from baseline in erosion index at the distal radius between the risedronate and placebo groups at Month 12 (the lower the percent change in erosion index, the greater the improvement of structural degradation); the last valid postbaseline measurement was to be used when the Month 12 value was missing (Last Observation Carried Forward or LOCF).
  NOTE: The study was unable to recruit sufficient numbers of patients to meet with the protocol specified numbers, thus it was terminated early after 5 months. No efficacy analyses were performed.
Time Frame: 12 months
Population: Study was terminated prior to acquiring any efficacy endpoints. No efficacy analyses were performed.
Arm/Group | One 150 mg Risedronate Once a Month | Placebo Tablet Once a Month
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Erosion Index of the Distal Radius
Description: Study was terminated prior to acquiring any efficacy endpoints. No efficacy analyses were performed.
Time Frame: 6 months
Population: Study was terminated prior to acquiring any efficacy endpoints. No efficacy analyses were performed.
Arm/Group | One 150 mg Risedronate Once a Month | Placebo Tablet Once a Month
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the point of study enrolment until the subject's last observation.
Description: Specific safety parameters and procedures were to include vital signs, serum chemistry panel/hematology/urinalysis, and recording of AEs, including moderate-to-severe upper GI events and clinical fractures.
Arm/Group | One 150 mg Risedronate Once a Month | Placebo Tablet Once a Month
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 2/7 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One 150 mg Risedronate Once a Month (N=7) | Placebo Tablet Once a Month (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngitis (General disorders) | 0 (0) | 1 (1)
Blood pressure increased (Cardiac disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
NOTE: The study was terminated early (after 5 months), prior to acquiring any efficacy endpoints; consequently, NO subject efficacy analyses were performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Site and Principal Investigator agree that all data, calculations, interpretations, opinions, and recommendations regarding the study will be the property of the Sponsor. The Study Site and Principal Investigator agree to consider the results as confidential information subject to use restrictions.

The names of the Investigator(s) will not be used by P&GP for commercial purposes without appropriate written permission, unless required by law or government regulation.